CLINICAL TRIAL: NCT02619695
Title: Comparison of Ketoprofen Gel to Placebo in Patients Presented With Mechanical Low Back Pain to the Emergency Department: A Randomized Placebo Controlled Trial
Brief Title: Comparison of Ketoprofen Gel to Placebo in Mechanical Low Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Collaborators: Pamukkale University (Other); Celal Bayar University (Other); Kocatepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015/08
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Low Back Pain
Keywords: ketoprofen; gel; low back pain; emergency department
MeSH Terms: conditions — Low Back Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketoprofen (Experimental): Interventional arm: ketoprofen gel 2.5% ketoprofen gel (Fastjel) has been administer as 2 gr in 5 cm area.
  Interventions: Drug: Fastjel
- Placebo (Placebo Comparator): Placebo arm: placebo gel form of ketoprofen
  Interventions: Drug: Fastjel

INTERVENTIONS:
Drug: Fastjel — 2.5% ketoprofen gel (Fastjel) has been administer as 2 gr in 5 cm area.

SUMMARY:
Mechanical low back pain is one most important emergency department presentations of patients seeking pain relief. Although parenteral pain killers such as opioids, non-steroidal anti-inflamatuar drugs and paracetamol are used commonly in these patients, application of analgesics in gel forms might be an reasonable alternative to these drugs with fewer adverse effects.

DETAILED DESCRIPTION:
Mechanical low back pain is one most important emergency department presentations of patients seeking pain relief. Parenteral pain killers such as opioids, non-steroidal anti-inflamatuar drugs (NSAID) and paracetamol are used commonly in these patients. However, these drugs are not out of adverse effects and can not be used in some patients with diverse comorbidities. Gel forms of NSAIDs are used commonly in the outpatient clinics and shown to be effective in these patients by a Cochrane meta-analysis. However, there is no data on the effect of gel forms of analgesics in ED. The application of analgesics in gel forms might be a reasonable alternative to the paranteral drugs with fewer adverse effects.

The present study aimed to reveal the effect of ketoprofen gel in patients presented with low back pain to emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical low back pain

Exclusion Criteria:

* Under 18 years old
* Over 65 years old
* Pain less than 40 mm in visual analogue scale
* Allergy to the study drug
* Drug or alcohol addiction
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale at 30 minutes | 30 minutes

SECONDARY OUTCOMES:
Adverse effects | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Serinken, Professor, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

REFERENCES:
- [Background] Friedman BW, Dym AA, Davitt M, Holden L, Solorzano C, Esses D, Bijur PE, Gallagher EJ. Naproxen With Cyclobenzaprine, Oxycodone/Acetaminophen, or Placebo for Treating Acute Low Back Pain: A Randomized Clinical Trial. JAMA. 2015 Oct 20;314(15):1572-80. doi: 10.1001/jama.2015.13043. PMID 26501533
- See also: Pubmed link — http://www.ncbi.nlm.nih.gov/pubmed/26501533